CLINICAL TRIAL: NCT03367624
Title: Epidemiology of Post-influenza Bacterial Pneumonia Due to a Panton-Valentine Leukocidin Positive Staphylococcus Aureus
Acronym: FLUVALENTINE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2017/FLUVALENTINE-BAUX/YB
Record Dates: First submitted 2017-11-18; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Influenza; Staphylococcus Aureus Pneumonia; PV Leukocidin
Keywords: influenza; Staphylococcus Aureus; Pneumonia; PV leukocidin; ICU
MeSH Terms: conditions — Influenza, Human; Pneumonia, Staphylococcal; Staphylococcal Infections; Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Secondary bacterial influenza pneumonia caused by Panton-Valentine Leukocidin Positive Staphylococcus aureus is a rare complication but with poor prognosis. This pathology seems to affect young patients (20-40 years) without any medical history. Since the influenza pandemic of 2009, this complication is more and more mentioned, sought and diagnosed. However, the literature is poor, consisting of case reports, experimental studies on murine models, and low-power studies.

The main objective is to evaluate the mortality in intensive care units of patients post-influenza bacterial pneumonia due to a Panton-Valentine Leukocidin positive Staphylococcus aureus

ELIGIBILITY:
Inclusion Criteria:

* Patient treated for post-influenza bacterial pneumonia due to a Panton-Valentine Leukocidin positive Staphylococcus aureus in intensive care unit

Exclusion Criteria:

* Minor patient
* Patient under protective measurement
* Absence of bacteriological and / or virological documentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care units for the management of influenza pneumonia infected with Panton-Valentine Leukocidin Positive Staphylococcus aureus over a retrospective period from 2009 to winter 2016-2017.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of dead patients | During Length of stay in intensive care unit (an average of 2 weeks)
  All cause of mortality

SECONDARY OUTCOMES:
Demographic data relating to age | Baseline
  age
Demographic data relating to sex | Baseline
  sex
Respiratory failure | Baseline
  PaO2/iFO2 value
Demographic data relating to immunosuppression | Baseline
  Amount of polynuclear neutrophils (G/L)
risk factors for methicillin-resistant Staphylococcus aureus | Baseline
  hospitalization
risk factors for methicillin-resistant Staphylococcus aureus | Baseline
  dialysis
risk factors for methicillin-resistant Staphylococcus aureus | Baseline
  surgery
risk factors for methicillin-resistant Staphylococcus aureus | Baseline
  presence of percutaneous or long-term catheter
Clinical data relating to pre-admission antibiotics | Baseline
  type of antibiotic prescribed
Clinical data in the initial phase relating to SAPS 2 score | Baseline
  Simplified acute Physiology score (SAPS2) score between 0 and 163 and a predicted mortality between 0% and 100%
Clinical data in the initial phase relating to SOFA admission | Baseline
  Sequential Organ Failure Assessment (SOFA)
Clinical data in the initial phase relating to neutropenia | During Length of stay in intensive care unit (an average of 2 weeks)
  neutropenia
Clinical data in the initial phase relating to neutropenia | During Length of stay in intensive care unit (an average of 2 weeks)
  thrombocytopenia
Clinical data in the initial phase relating to metabolic acidosis | During Length of stay in intensive care unit (an average of 2 weeks)
  metabolic acidosis
Clinical data in the initial phase relating to oxygen dependence | During Length of stay in intensive care unit (an average of 2 weeks)
  oxygen dependence
Clinical data in the initial phase relating to hyperthermia | During Length of stay in intensive care unit (an average of 2 weeks)
  hyperthermia
Clinical data in the initial phase relating to chills | During Length of stay in intensive care unit (an average of 2 weeks)
  chills
Clinical data in the initial phase relating to headhache | During Length of stay in intensive care unit (an average of 2 weeks)
  headache
Clinical data in the initial phase relating to productive cough | During Length of stay in intensive care unit (an average of 2 weeks)
  productive cough
Clinical data in the initial phase relating to dyspnoea | During Length of stay in intensive care unit (an average of 2 weeks)
  dyspnoea
Clinical data in the initial phase relating to acute respiratory failure | During Length of stay in intensive care unit (an average of 2 weeks)
  acute respiratory failure
Clinical data in the initial phase relating to hemoptysis | During Length of stay in intensive care unit (an average of 2 weeks)
  hemoptysis
Clinical data in the initial phase relating to uni - or multi - lobar infiltration on chest X - ray or CT scan | During Length of stay in intensive care unit (an average of 2 weeks)
  uni - or multi - lobar infiltration on chest X - ray or CT scan
Clinical data in the initial phase relating to pleural effusion | During Length of stay in intensive care unit (an average of 2 weeks)
  pleural effusion
Clinical data in the initial phase | During Length of stay in intensive care unit (an average of 2 weeks)
  necrotizing pneumonitis
Clinical data in the initial phase relating to renal failure | During Length of stay in intensive care unit (an average of 2 weeks)
  renal failure according to KDIGO classification
Prognostic factors for this pathology | During Length of stay in intensive care unit (an average of 2 weeks)
  Time to diagnosis of influenza infection and Panton-Valentine Leukocidin Positive Staphylococcus aureus Haemoptysis, leukopenia, thrombocytopenia, acute respiratory distress syndrome (ARDS), PaO2 / Fi02, inotropic support
Complications | During Length of stay in intensive care unit (an average of 2 weeks)
  Complications related to Septic shock ARDS: according to Berlin 2009 classification Extra corporeal vein-venous or veino-arterial oxygenation membrane (ECMO VV or ECMO VA) Ischemic limb Pneumothorax Acute renal failure according to Kdigo classification Disseminated intravascular coagulation (DIC) (2) Cardiogenic shock / cardiogenic pulmonary acute edema Multi visceral failure syndrome (3) Use of surgery: abscess drainage, lobectomy, amputation, laparotomy and colonic resection ...
Collection of infectious samples | During Length of stay in intensive care unit (an average of 2 weeks)
  Bacteriological, Parasitological, Virological
Probabilistic antibiotherapy | During Length of stay in intensive care unit (an average of 2 weeks)
  Collection of probabilistic antibiotherapy
Probabilistic antibiotherapy | During Length of stay in intensive care unit (an average of 2 weeks)
  Duration of probabilistic antibiotherapy
Prescribed antibiotic therapy | During Length of stay in intensive care unit (an average of 2 weeks)
  Collection of Prescribed antibiotic therapy
Prescribed antibiotic therapy | During Length of stay in intensive care unit (an average of 2 weeks)
  Duration for the appropriate anti-toxin treatment
Collection of the date of introduction of adapted antibiotic therapy | During Length of stay in intensive care unit (an average of 2 weeks)
  Collection of the date of introduction of adapted antibiotic therapy
Number of patients with Influenza type A | During Length of stay in intensive care unit (an average of 2 weeks)
  Number of patients with Influenza type A
Number of patients with Influenza type B | During Length of stay in intensive care unit (an average of 2 weeks)
  Number of patients with Influenza type B
Date of initiation of anti-viral treatment in relation to the onset of symptoms and duration of anti-viral treatment | During Length of stay in intensive care unit (an average of 2 weeks)
  Date of initiation of anti-viral treatment in relation to the onset of symptoms and duration of anti-viral treatment
Dosage of antiviral treatment | During Length of stay in intensive care unit (an average of 2 weeks)
  Dosage of antiviral treatment
Number of serious influenza infections per year and per center with early and late deaths | During Length of stay in intensive care unit (an average of 2 weeks)
  Mortality caused by serious inflenza infections

CONTACTS AND LOCATIONS:
Locations (1):
- Baux, Nancy, France